CLINICAL TRIAL: NCT00940329
Title: Investigation on the Cardiovascular and Pharmacokinetic Interaction Between Oral Roflumilast and Inhaled Formoterol in Healthy Subjects
Brief Title: Pharmacodynamic/Pharmacokinetic Interactions Between Oral Roflumilast and Inhaled Formoterol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BY217/CP-059
Record Dates: First submitted 2009-07-03; First posted 2009-07-16 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: Drug interactions; Pharmacodynamic interactions; Pharmacokinetic interactions; Formoterol; Healthy subjects; Phase I study; Roflumilast
MeSH Terms: interventions — Roflumilast

ARMS (2):
- Treatment A (Active Comparator)
  Interventions: Drug: Roflumilast
- Treatment B (Active Comparator)
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: Roflumilast — Treatment A (500 μg/d roflumilast from day 2 to day 18 and 48 μg/d formoterol from day 12 to day 18)
  Arms: Treatment A
Drug: Roflumilast — Treatment B (48 μg/d formoterol from day 2 to day 18 and 500 μg/d roflumilast from day 9 to day 18)
  Arms: Treatment B

SUMMARY:
This Phase I, open, randomized controlled, multiple-dose, parallel-group study investigated the potential pharmacodynamic and pharmacokinetic interactions between multiple doses of oral roflumilast and inhaled formoterol. Healthy male subjects were assigned to treatment A or treatment B. Subjects in treatment A received 500 μg/d roflumilast from day 2 to day 18 and 48 μg/d formoterol from day 12 to day 18. Subjects in treatment B received 48 μg/d formoterol from day 2 to day 18 and 500 μg/d roflumilast from day 9 to day 18. Impedance cardiography, ECG, serum potassium and glucose concentrations and effects on blood eosinophils assessed potential pharmacodynamic interactions. In addition, the safety and tolerability were evaluated. Pharmacokinetic parameters were assessed for roflumilast, roflumilast N-oxide, and formoterol.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Normal body weight as indicated by a Body Mass Index (BMI) between 18 and 30 kg/m2 and a body weight > 50 kg
* Assessed as healthy, based on a screening examination including medical history, physical examination, BP, PuR, ECG, and clinical laboratory results
* Caucasian

Exclusion Criteria:

* Suspected lack of compliance
* Participant in any other study or donation of blood during the last 30 d before start of this study (last day of intake of medication - first day of medication in the following study)
* Any active disease, acute or chronic (also psychiatric diseases)
* Any signs or present history of cardiac diseases (e.g. QTc interval acc. to Bazett ≥ 430 ms, PQ ≥ 220 ms), in particular tachycardiac arrhythmia, third-degree AV-block, idiopathic-subvalvular aortic stenosis or hypertrophic-obstructive cardiomyopathia
* Proneness to symptomatic orthostatic dysregulation, fainting or "blackouts" (medical history), or to orthostatic hypotension defined by SBP < 90 mm Hg (standing blood pressure, 30 s after raising up from a supine position)
* Gastrointestinal surgery except from appendectomy and herniotomy
* HIV or hepatitis screening positive or not performed (in case of a positive HIV test, the subject had to be informed by a physician in personal communication
* Drug screening positive or not performed
* Excessive xanthine consumption (more than 5 cups of coffee or equivalent per day)
* Non-compliance for measurements of impedance cardiography (feasibility was proven and documented at the screening visit by one test procedure)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2004-04; Primary Completion 2004-07 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Potential cardiovascular interaction (exploratory)

SECONDARY OUTCOMES:
Potential pharmacokinetic interactions and potential pharmacodynamic interactions
Safety and tolerability of the monotreatments and the combination treatment (exploratory)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Nycomed, Konstanz, Germany

REFERENCES:
- [Derived] de Mey C, Nassr N, Lahu G. No relevant cardiac, pharmacokinetic or safety interactions between roflumilast and inhaled formoterol in healthy subjects: an open-label, randomised, actively controlled study. BMC Clin Pharmacol. 2011 Jun 1;11:7. doi: 10.1186/1472-6904-11-7. PMID 21631929
- See also: BY217-CP-059-RDS-2005-05-03.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4469&filename=BY217-CP-059-RDS-2005-05-03.pdf